CLINICAL TRIAL: NCT07283289
Title: Prospective Observational Cohort Study on the Prevalence of Obstructive Sleep Apnea in Patients With Peripheral Arterial Occlusive Disease
Brief Title: Prevalence of Obstructive Sleep Apnea in Patients With Peripheral Arterial Occlusive Disease
Acronym: OSAPAD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-014
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Artery Disease
Keywords: Obstructive Sleep Apnea Syndrome; Polygraphy; Diagnosis; Prevalence; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Sleep Apnea, Obstructive; Disease; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PAOD: Patients hospitalized or seen in vascular medicine consultation with a diagnosis of PAOD at all stages (operated or not) according to the Leriche and Fontaine classification.

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is characterized by partial (hypopnea) or complete (apnea) obstruction of the upper airways, leading to intermittent hypoxemia and sleep fragmentation. Peripheral arterial occlusive disease (PAOD) is a chronic condition defined by the narrowing or occlusion of arteries in the lower limbs, often resulting in ischemia of downstream tissues. This disease is a common complication of atherosclerosis and affects approximately 1.2% of the general French population.

OSAS is a well-established risk factor for atherosclerotic disease, particularly for coronary and neurovascular events. Although a relationship between OSAS and PAOD has been investigated in recent years, the link has not been definitively established and requires further study. Therefore, this preliminary cohort study aims to observe the prevalence of OSAS among patients diagnosed with PAOD, regardless of the disease stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with a confirmed diagnosis of PAOD, seen either during hospitalization or in an outpatient vascular medicine consultation. Inclusion is permitted regardless of the disease stage (according to the Leriche and Fontaine classification) or prior surgical intervention.
3. No objection to the use of their pseudonymised medical data
4. Polygraphy scheduled as part of routine care within one month.

Exclusion Criteria:

1. Inability to perform the Ankle-Brachial Index (ABI) or sleep polygraphy due to physical or cognitive constraints (e.g., severe dementia, limb malformation, etc.).
2. History of OSAS diagnosis confirmed by polygraphy, and currently receiving nocturnal treatment (e.g., Continuous Positive Airway Pressure - CPAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of PAOD, seen either during hospitalization or in an outpatient vascular medicine consultation.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with OSAS | Up to 1 month
  Patients diagnosed with OSAS by polygraphy, regardless of severity.

SECONDARY OUTCOMES:
Proportion of patients diagnosed with OSAS, stratified by the presence or absence of cardiovascular comorbidities. | Up to 1 month
  The prevalence of OSAS will be analyzed in patients with PAOD, stratified by the presence or absence of cardiovascular involvement (e.g., carotid plaque, carotid stenosis, or abdominal aortic aneurysm).
Ankle-brachial index | Day 0
  The Ankle-Brachial Index (ABI) will be analyzed according to OSAS severity, which is defined by the Apnea-Hypopnea Index (AHI):
  * Mild: 5 to 14 events per hour
  * Moderate: 15 to 30 events per hour
  * Severe: > 30 events per hour
Toe-brachial index | Day 0
  The toe-Brachial Index (TBI) will be analyzed according to OSAS severity, which is defined by the Apnea-Hypopnea Index (AHI):
  * Mild: 5 to 14 events per hour
  * Moderate: 15 to 30 events per hour
  * Severe: > 30 events per hour
Proportion of patients diagnosed with OSAS according to PAOD severity | Up to 1 month
  The prevalence of OSAS (diagnosed by polygraphy) will be analyzed according to the severity stage of PAOD.

CONTACTS AND LOCATIONS:
Overall Officials: Léonie GEY, M.D., Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No